CLINICAL TRIAL: NCT00715078
Title: A Randomized, Multicenter, Single Blind Study in Men With Metastatic Androgen Independent Prostate Cancer to Evaluate Sipuleucel-T Manufactured With Different Concentrations of PA2024 Antigen
Brief Title: To Evaluate Sipuleucel-T Manufactured With Different Concentrations of (PA2024) Antigen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dendreon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P07-2
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-04

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostate; immune therapy; immunotherapy; vaccine; dendritic cells; antigen-presenting cells; antigen presenting cells; cancer vaccine; prostate specific antigen (PSA); prostatic adenocarcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sipuleucel-T

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A (Active Comparator): Sipuleucel-T with the concentration of 10 μg/mL PA2024 in a cell suspension of 1 x 10^7 peripheral blood mononuclear cells (PBMCs) per mL. Subjects received infusion of sipuleucel-T, at 2-week intervals, for a total of 3 infusions.
  Interventions: Biological: sipuleucel-T
- Cohort B (Active Comparator): Sipuleucel-T with the concentration of 5 μg/mL PA2024 in a cell suspension of 1 x 10^7 PBMCs per mL. Subjects received infusion of sipuleucel-T, at 2-week intervals, for a total of 3 infusions.
  Interventions: Biological: sipuleucel-T
- Cohort C (Active Comparator): Sipuleucel-T with the concentration of 2 μg/mL PA2024 in a cell suspension of 1 x 10^7 PBMCs per mL. Subjects received infusion of sipuleucel-T, at 2-week intervals, for a total of 3 infusions.
  Interventions: Biological: sipuleucel-T

INTERVENTIONS:
Biological: sipuleucel-T — Sipuleucel-T is an autologous cellular product consisting of antigen presenting cells (APCs) activated with PA2024, a recombinant fusion protein composed of prostatic acid phosphatase (PAP), linked to granulocyte-macrophage colony-stimulating factor (GM-CSF)

SUMMARY:
This is a randomized, multicenter, single blind, Phase 2 trial of immunotherapy in men with metastatic androgen independent prostate cancer to evaluate sipuleucel-T manufactured with different concentrations of PA2024 antigen

DETAILED DESCRIPTION:
This is a randomized, multicenter, single blind, Phase 2 trial of immunotherapy in men with metastatic androgen independent prostate cancer to evaluate sipuleucel-T manufactured with 1 of 3 different concentrations of PA2024 antigen The primary purpose of this study is to compare the changes in CD54 upregulation between each of these 3 groups of subjects.

ELIGIBILITY:
Inclusion Criteria:

For a subject to be eligible for participation in this study, all of the following criteria must be satisfied.

* Histologically documented adenocarcinoma of the prostate.
* Metastatic disease.
* Progressive androgen independent castrate resistant prostate cancer.
* Serum PSA ≥ 5.0 ng/mL.
* Life expectancy of ≥ 6 months.
* Castrate level of testosterone (< 50 ng/dL) achieved via medical or surgical castration.
* Men ≥ 18 years of age.
* Adequate hematologic, renal and liver function.

Exclusion Criteria:

A subject will not be eligible for participation in this study if any of the following criteria apply.

* The presence of known lung, liver, or brain metastases, malignant pleural effusions, or malignant ascites.
* A requirement for treatment with opioid analgesics for any reason within 21 days prior to registration.
* Moderate to severe disease related pain.
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2.
* Use of non-steroidal antiandrogens within 6 weeks of registration.
* Anti-androgen withdrawal response.
* Treatment with chemotherapy within 3 months of registration.
* More than 2 chemotherapy regimens prior to registration.
* Initiation or discontinuation of bisphosphonate therapy within 28 days prior to registration.
* Treatment with any of the following medications or interventions within 28 days of registration:

  * Systemic corticosteroids,
  * External beam radiation therapy or surgery,
  * Dietary and herbal supplements, as well as alternative treatments that have evidence of hormonal and/or anticancer properties (e.g., prostate cancer (PC) -SPES or PC-SPEC) and saw palmetto,
  * Megestrol acetate (Megace®), diethylstilbesterol (DES), or cyproterone acetate, ++Ketoconazole,
  * 5-alpha-reductase inhibitors,
  * High dose calcitriol [1,25(OH)2Vitamin D] (i.e., > 0.5 mcg/day).
* Any other systemic therapy for prostate cancer (except for medical castration).
* Treatment with any investigational vaccine within 2 years of registration or treatment with any other investigational product within 28 days of registration.
* Participation in any previous study involving sipuleucel-T, regardless of whether the subject received sipuleucel-T (APC8015) or placebo.
* Known pathologic long-bone fractures, imminent pathologic long-bone fracture (cortical erosion on radiography > 50%) or spinal cord compression.
* A history of stage III or greater cancer, excluding prostate cancer. Basal or squamous cell skin cancers must have been adequately treated and the subject must be disease-free at the time of registration. Subjects with a history of stage I or II cancer must have been adequately treated and been disease-free for ≥ 3 years at the time of registration.
* A requirement for systemic immunosuppressive therapy for any reason.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to sipuleucel-T or granulocyte-macrophage colony-stimulating factor.
* Any infection requiring parenteral antibiotic therapy or causing fever (temp > 100.5°F or > 38.1°C) within 1 week prior to registration.
* Any medical intervention or other condition which, in the opinion of the Principal Investigator or the Dendreon Medical Monitor, could compromise adherence with study requirements or otherwise compromise the study's objectives.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Israel, MD, Study Director — Valeant Pharmaceuticals North America LLC
Locations (12):
- United States (12):
  - UCSD Moores Cancer Center, La Jolla, California
  - Sharp Clinical Oncology Research, San Diego, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Indiana University, Indianapolis, Indiana
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Providence Medical Center, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Northwest Cancer Specialists, Portland, Oregon
  - Urology of Virginia, Sentara Medical Group, Norfolk, Virginia
  - Virginia Mason Medical Center Urology and Renal Transplantation, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: National Alliance of State Prostate Cancer Coalitions — http://www.naspcc.org
- See also: Us TOO International — http://www.ustoo.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Sipuleucel-T with the concentration of 10 μg/mL PA2024 in a cell suspension of 1 x 10^7 PBMCs per mL. Subjects received infusion of sipuleucel-T, at 2-week intervals, for a total of 3 infusions.
Period: Overall Study
Arm/Group | Cohort A | Cohort B | Cohort C
Started | 41 | 40 | 41
Received ≥ 1 Study Infusion | 40 | 40 | 39
Received ≥ 1 Leukapheresis | 40 | 40 | 40
Completed | 11 | 4 | 3
Not Completed | 30 | 36 | 38
Not completed — Death | 29 | 36 | 36
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Unable to start due to disease prog. | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B | Cohort C | Total
Number analyzed (Participants) | 41 | 40 | 41 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 9 | 11 | 31
  >=65 years | 30 | 31 | 30 | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (8.25) | 71.8 (8.29) | 68.6 (7.5) | 70.5 (8.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 41 | 40 | 41 | 122
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 3 | 6
  White | 38 | 35 | 38 | 111
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 41 | 40 | 41 | 122
Eastern Cooperative Oncology Group (ECOG) performance status [Count of Participants; unit: Participants] — ECOG Performance Status is a method used to assess the functional status of a patient. The scale ranges from 0-5. 0=Fully active, able to carry on all pre-disease performance without restriction; 1=Restricted in physically strenuous activity but ambulatory and able to carry out light or sedentary work; 2=Ambulatory, capable of all self-care but unable to carry out work activities. Up and about >50% of waking hour; 3=Capable of limited self-care, confined to bed or chair >50% of waking hours; 4=Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; 5=Dead
  Participants
    ECOG 0=Fully Active; No restrictions | 29 | 24 | 27 | 80
    ECOG 1= Restricted Strenuous Activity | 12 | 16 | 14 | 42
Gleason Score [Count of Participants; unit: Participants] — Gleason score= prostate cancer grading system based on how tissue looks under a microscope. Scores range 2-10 and indicates how likely it is that a tumor will spread. A low score means the cancer tissue is similar to normal tissue and the tumor is less likely to spread. Gleason Score ≤ 6=the tumor is well differentiated, less aggressive and likely to grow more slowly;7=the tumor is moderately differentiated, moderately aggressive, and likely to grow but may not spread quickly;≥8=the tumor is poorly differentiated or undifferentiated, highly aggressive, and likely to grow faster and spread.
  Participants
    Gleason Score ≤ 6 | 7 | 8 | 4 | 19
    Gleason Score =7 | 12 | 15 | 14 | 41
    Gleason Score ≥ 8 | 22 | 16 | 23 | 61
    Missing information | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Cumulative CD54 Upregulation Ratio Between Each of the Cohorts.
Description: An analysis of variance model for the log transformed cumulative CD54 upregulation ratio (CD54 upregulation is the fold increase in the final product (FP) from buoyant density separations (BDS) step 65. BDS65 step refers to sample taken after both BDS77 and BDS65 but before ex vivo culture in the presence of antigen PA2024. FP refers to sample taken after ex vivo culture) that includes the antigen concentration cohort as the independent variable was performed. Subjects who received all 3 infusions were included.
Time Frame: Baseline, Months 2, 4 and 6.
Population: Cumulative CD54 upregulation ratio will be the primary end point and calculated as the sum of Infusion 1 through Infusion 3 final product values for each infused subject.
Measure: Mean (Standard Error); unit: Ratio ofCD54 molecules on BDS65:FP cells
Arm/Group | Cohort A | Cohort B | Cohort C
Number analyzed (Participants) | 40 | 36 | 37
Ratio ofCD54 molecules on BDS65:FP cells | 29.53 (1.285) | 30.94 (1.418) | 26.67 (1.194)
Statistical Analysis 1: Comparison: Cohort A vs Cohort B; The sample size determination is based on a standard deviation of 0.45 for the log transformed CD54 upregulation ratio estimated from previous studies assuming there is no difference in central values between the two compared cohorts. A sample size of 38 subjects per cohort will provide 70% power for the non-inferiority test for the two pairwise comparisons (Cohort B vs. Cohort A and Cohort C vs. Cohort A); Test type: Non-Inferiority or Equivalence — Cohort B is considered non-inferior to Cohort A if the lower limit of the 90% confidence interval (CI) for the ratio of Cohort B vs. Cohort A in the geometric mean of cumulative CD54 upregulation ratio is >0.8. The use of one-sided CI is based on an assumption that a higher concentration will correspond to a higher CD54 upregulation ratio. The use of 0.8 as margin is based on the assumption that a relative difference of <20% in upregulation ratios may not be clinically significant; p = 0.5019, ANOVA; ratio of geometric means (GeoMean) = 1.046, 90% CI 2-sided [0.936 to 1.168]
Statistical Analysis 2: Comparison: Cohort A vs Cohort C; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — Cohort C is considered non-inferior to Cohort A if the lower limit of the 90% confidence interval for the ratio of Cohort C vs. Cohort A in the geometric mean of cumulative CD54 upregulation ratio is >0.8. The use of one-sided CI is based on an assumption that a higher concentration will correspond to a higher CD54 upregulation ratio. The use of 0.8 as margin is based on the assumption that a relative difference of <20% in upregulation ratios may not be clinically significant; p = 0.1443, ANOVA; the ratio of geometric means = 0.907, 90% CI 2-sided [0.813 to 1.013]

ADVERSE EVENTS:
Time Frame: Baseline visit and at each visit through Month 6, or the initiation of an anticancer intervention, whichever occurs first.
Description: Following Month 6 (or the initiation of an anticancer intervention), treatment-related adverse events will be collected until death. All cerebrovascular events occurring throughout the study (regardless of causality) were reported. Adverse events are reported in the safety population defined as subjects that received ≥ 1 leukapheresis.
Groups:
- Cohort A: Sipuleucel-T with the concentration of 10 μg/mL PA2024 in a cell suspension of 1 x 10^7 peripheral blood mononuclear cells (PBMCs) per mL
- Cohort B: Sipuleucel-T with the concentration of 5 μg/mL PA2024 in a cell suspension of 1 x 10^7 PBMCs per mL
- Cohort C: Sipuleucel-T with the concentration of 2 μg/mL PA2024 in a cell suspension of 1 x 10^7 PBMCs per mL
Arm/Group | Cohort A | Cohort B | Cohort C
All-Cause Mortality (participants affected / at risk) | 29/40 | 36/40 | 36/40
Serious Adverse Events (participants affected / at risk) | 10/40 | 9/40 | 11/40
Other Adverse Events (participants affected / at risk) | 38/40 | 40/40 | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=40) | Cohort B (N=40) | Cohort C (N=40)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 0 (0)
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ATRIOVENTRICULAR BLOCK SECOND DEGREE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
BRADYCARDIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
ASTHENIA (General disorders) | 3 (3) | 1 (1) | 0 (0)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0)
DISEASE PROGRESSION (General disorders) | 1 (1) | 1 (1) | 1 (1)
FATIGUE (General disorders) | 0 (0) | 1 (1) | 2 (2)
NON-CARDIAC CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 1 (1) | 0 (0)
BACTERAEMIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
WOUND (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
INTRACRANIAL TUMOUR HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
BLADDER OUTLET OBSTRUCTION (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
URETHRAL STENOSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A (N=40) | Cohort B (N=40) | Cohort C (N=40)
ANAEMIA (Blood and lymphatic system disorders) | 6 (6) | 4 (5) | 8 (8)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 (4) | 2 (3) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 9 (10) | 8 (9) | 6 (7)
DIARRHOEA (Gastrointestinal disorders) | 4 (5) | 4 (4) | 3 (3)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
FLATULENCE (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 16 (20) | 11 (11) | 11 (12)
RETCHING (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 8 (9) | 5 (5) | 5 (6)
ASTHENIA (General disorders) | 2 (2) | 3 (3) | 4 (5)
CHEST DISCOMFORT (General disorders) | 0 (0) | 1 (1) | 2 (2)
CHEST PAIN (General disorders) | 6 (6) | 0 (0) | 2 (2)
CHILLS (General disorders) | 9 (15) | 13 (25) | 10 (15)
FATIGUE (General disorders) | 20 (23) | 20 (27) | 16 (17)
INFLUENZA LIKE ILLNESS (General disorders) | 4 (6) | 0 (0) | 4 (6)
MALAISE (General disorders) | 1 (2) | 0 (0) | 2 (2)
OEDEMA PERIPHERAL (General disorders) | 6 (6) | 9 (10) | 4 (5)
PAIN (General disorders) | 0 (0) | 4 (6) | 1 (1)
PYREXIA (General disorders) | 5 (6) | 4 (5) | 7 (8)
BRONCHITIS (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
GASTROENTERITIS VIRAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 3 (3) | 1 (1)
PNEUMONIA (Infections and infestations) | 0 (0) | 2 (2) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (3) | 2 (2) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 5 (6) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
CITRATE TOXICITY (Injury, poisoning and procedural complications) | 5 (10) | 4 (7) | 6 (13)
CONTUSION (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (4)
LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (3)
BLOOD PRESSURE INCREASED (Investigations) | 2 (2) | 1 (1) | 2 (7)
WEIGHT DECREASED (Investigations) | 7 (7) | 5 (5) | 3 (3)
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 (8) | 10 (10) | 8 (8)
DEHYDRATION (Metabolism and nutrition disorders) | 8 (12) | 4 (8) | 4 (6)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 (16) | 13 (19) | 7 (13)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 10 (15) | 16 (21) | 12 (16)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 5 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5) | 4 (4) | 1 (1)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (7) | 2 (2)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 1 (1)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 8 (9) | 4 (5) | 12 (13)
MYALGIA (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (5) | 4 (5)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 6 (8) | 3 (6) | 9 (9)
DIZZINESS (Nervous system disorders) | 6 (7) | 6 (6) | 8 (11)
DYSGEUSIA (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 4 (5) | 3 (3) | 7 (8)
HYPOAESTHESIA (Nervous system disorders) | 1 (1) | 5 (11) | 1 (1)
PARAESTHESIA (Nervous system disorders) | 3 (3) | 9 (12) | 5 (5)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 2 (3) | 2 (3)
SOMNOLENCE (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
TREMOR (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
AGITATION (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2)
ANXIETY (Psychiatric disorders) | 3 (4) | 6 (7) | 3 (3)
DEPRESSION (Psychiatric disorders) | 5 (5) | 1 (1) | 3 (3)
INSOMNIA (Psychiatric disorders) | 3 (3) | 5 (5) | 6 (6)
HAEMATURIA (Renal and urinary disorders) | 5 (6) | 4 (6) | 1 (1)
HYDRONEPHROSIS (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
NOCTURIA (Renal and urinary disorders) | 2 (2) | 5 (5) | 2 (2)
POLLAKIURIA (Renal and urinary disorders) | 1 (1) | 4 (4) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 3 (3) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2) | 3 (3)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (3)
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
HAEMATOMA (Vascular disorders) | 3 (3) | 2 (2) | 0 (0)
HOT FLUSH (Vascular disorders) | 1 (1) | 1 (1) | 2 (3)
HYPERTENSION (Vascular disorders) | 3 (6) | 4 (5) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 4 (4)
PARAESTHESIA ORAL (Gastrointestinal disorders) | 2 (4) | 3 (5) | 5 (9)
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 3 (3) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the Study will be published and/or presented in an integrated manner reflecting the results observed across all participating centers. Accordingly, decisions on timing and content of publications and presentations relating to the Study will be coordinated by Dendreon in communication with institutions contributing patients to the Study.